CLINICAL TRIAL: NCT02444871
Title: Immunoglobulin-M-enriched (IgM-enriched) Immunoglobulin Attenuates Systemic Endotoxin Activity in Early Severe Sepsis
Brief Title: IgM-enriched Immunoglobulin Attenuates Systemic Endotoxin Activity in Early Severe Sepsis
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Saskia Wand, Dr. Saskia Wand, Goethe University
Other Study IDs: DEEP Trial
Record Dates: First submitted 2015-05-09; First posted 2015-05-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Sepsis
Keywords: IgM-enriched immunoglobulins; endotoxin activity assay; thrombelastometry; aggregometry
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effect of IgM-enriched immunoglobulins (Pentaglobin) on the endotoxin activity, conventional coagulation parameters, viscoelastic and aggregometric measurements of patients with severe sepsis.

DETAILED DESCRIPTION:
Before the change of the standard operating procedure (SOP) with the implementation of the application of IgM-enriched immunoglobulins to patients with severe sepsis and septic shock conventional inflammatory and coagulation parameters, viscoelastic and aggregometric measurements as well as the endotoxin activity was measured in 15 patients. After the change of SOP the same parameters were recorded for additional 15 patients.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* proven or suspected severe sepsis or septic shock
* written consent of the patient or a legal person in charge

Exclusion Criteria:

* Pregnancy
* anticoagulation other than heparin
* Inherited coagulopathy or thrombophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis or septic shock in a surgical, tertiary care ICU
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in endotoxin activity | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  The endotoxin activity of the patients was measured with a point of care assay and noted in on an arbitrary scale from 0 to 1.0

SECONDARY OUTCOMES:
Changes in CT-NATEM | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Changes in clotting time (CT) of the naturally activated rotational thrombelastometry (ROTEM), results were noted in seconds.
Changes in MCF-NATEM | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Changes in maximum clot firmness (MCF) of the naturally activated rotational thrombelastometry (ROTEM), results were noted in millimeters.
Changes in CFT-NATEM | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Changes in clot formation time (CFT) of the naturally activated rotational thrombelastometry (ROTEM), results were noted in seconds.
Changes in NATEM-Alpha angle | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Changes in Alpha angle of the naturally activated rotational thrombelastometry (ROTEM), results were noted in °.
Changes in ADPtest | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Platelet activation was measured as the area under the curve of a multiple electrode aggregometry. Platelets were activated using adenosine diphosphate (ADPtest)
Changes in ASPItest | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Platelet activation was measured as the area under the curve of a multiple electrode aggregometry. Platelets were activated using arachidonic acid (ASPItest)
Changes in TRAPtest | Baseline, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78 and 84 hours
  Platelet activation was measured as the area under the curve of a multiple electrode aggregometry. Platelets were activated using thrombin receptor activating peptide (TRAPtest)
Platelet count | Baseline, 12, 24, 36, 48, 60, 72 and 84 hours
  Platelet count was determined in the clinical routine and noted /nl.
Interleukin-6 | Baseline, 12, 24, 36, 48, 60, 72 and 84 hours
  Interleukin-6 level was determined in the clinical routine and was noted in pg/ml.
Leukocyte count | Baseline, 12, 24, 36, 48, 60, 72 and 84 hours
  Leukocyte count was determined in the clinical routine and was noted /µl.
Lipopolysaccharide-binding-protein (LBP) | Baseline, 24, 48 and 72 hours
  Lipopolysaccharide-binding-protein (LBP) was determined in the clinical routine and was noted in µg/l.

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Wand S, Klages M, Kirbach C, Warszawska J, Meybohm P, Zacharowski K, Koch A. IgM-Enriched Immunoglobulin Attenuates Systemic Endotoxin Activity in Early Severe Sepsis: A Before-After Cohort Study. PLoS One. 2016 Aug 9;11(8):e0160907. doi: 10.1371/journal.pone.0160907. eCollection 2016. PMID 27504630